CLINICAL TRIAL: NCT05233748
Title: Neuromotor Control During Walking in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1125634
Record Dates: First submitted 2021-10-14; First posted 2022-02-10 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Cerebral Palsy
Keywords: locomotor control; balance
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Cross sectional study of responses to visual perturbations in two groups, children with CP and age-and sex- matched TD (typical development). Each group will undergo two stimulation conditions, stochastic resonance (SR) stimulation and a control / no stochastic resonance (noSR) condition while walking with and without visual perturbations.
Who Masked: Participant
Masking Description: The SRopt and noSR conditions will be presented in random order generated by a computer program and the subjects will be blinded to either condition, due to SR stimulation being below the sensory threshold i.e subjects do not perceive the stimulation at all.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stochastic Resonance (SR) (Experimental): During this condition, participants will walk on the treadmill while receiving SR stimulation at their individual optimal intensity (SR) with and without visual perturbations.
  Interventions: Device: Stochastic Resonance (SR)
- No Stochastic Resonance (noSR) (No Intervention): During this condition, participants will walk on the treadmill while receiving no SR stimulation (noSR) with and without visual perturbations.

INTERVENTIONS:
Device: Stochastic Resonance (SR) — The system consists of six linear isolated stimulators (STMISOLA, Biopac Systems, Inc., Goleta, USA). The SR signal (Gaussian White Noise, zero mean) will be generated through a 16 bit PCI 6733 National Instruments multifunction data acquisition card by a custom LabView program. The stimulation sites include the ankle, lateral soleus, peroneus longus, and tibialis anterior muscles and the hip.
  Arms: Stochastic Resonance (SR)

SUMMARY:
One out of every three children with cerebral palsy (CP) falls daily, with more than half of the falls occurring while walking. To avoid falling, the nervous system must continuously monitor how the body moves and, when an imbalance is detected, activate muscles for an appropriate correction. In this project, we will use small electrical stimulation of muscles and tendons that enhances the sense of body positioning, to allow children with CP to generate more accurate balance corrections.

ELIGIBILITY:
Inclusion Criteria:

* Age 8 - 24 years
* Diagnosis of spastic diplegic or hemiplegic CP (for participants with CP group only)
* GMFCS classification level I or II (ability to walk independently with using any assistive device)
* Visual, perceptual, and cognitive/ communication skills to follow multiple step commands
* Seizure-free or well controlled seizures
* Ability to communicate pain or discomfort during testing procedures
* Parental/guardian consent and child assent/consent

Exclusion Criteria:

* Diagnosis of athetoid, ataxic or quadriplegic CP
* Significant scoliosis (scoliometer angle > 9°)
* History of selective dorsal root rhizotomy
* Botox injections in the lower limb within the past 6 months
* Severe spasticity of the lower extremity muscles (e.g. a score of 4 on the Modified Ashworth Scale)
* Severely limited range of motion/ irreversible muscle contractures
* Lower extremity surgery or fractures in the year prior testing
* Joint instability or dislocation in the lower extremities
* Marked visual or hearing deficits

Ages: 8 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Change in Margin of Stability(MOS) | At the end of the session after 6 minutes of stimulation i.e Pre stimulation MOS - Post stimulation MOS.
  MOS refers to the distance between extrapolated center of mass (which includes center of mass position and velocity) and the base of support. It has been previously used to measure balance in children with cerebral palsy, patients with stroke, Parkinson Disease, and Multiple Sclerosis. We will measure center of mass using kinetics and kinematic computed through a motion capture system(Qualysis).
  For the visual perturbation conditions, we will use center of mass excursion as the primary outcome measure (since it has been used in prior studies in children and adults using visual perturbation protocols).

CONTACTS AND LOCATIONS:
Overall Officials: John Jeka, PhD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Undecided